CLINICAL TRIAL: NCT01532947
Title: Survival of Endodontically Treated and Restored Premolars: A Randomized Controlled Trial
Brief Title: Randomized Controlled Trial of Fiber Post Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Prof. Marco Ferrari, Professor, University of Siena
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: RCTFP1
Record Dates: First submitted 2012-02-05; First posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Restoration Survival

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- post restoration (Experimental)
  Interventions: Procedure: post placement
- no post restoration (No Intervention): no post placement

INTERVENTIONS:
Procedure: post placement — placement of an endocanalar post
  Other Names: Prefabricated post DT LightPost, RTD; Customized post, EverStick Post, StickTech
  Arms: post restoration

SUMMARY:
This in vivo study examined the contribution of remaining coronal dentin and placement of a prefabricated or customized fiber post to the six-year survival of endodontically treated premolars. A sample of 345 patients provided 6 groups of 60 premolars in need of endodontic treatment. Groups were classified according to the number of remaining coronal walls before abutment build-up. Within each group, teeth were allocated to three subgroups: A) no post-retention; B) LP; C) ES (N=20). All teeth were protected with a crown. Cox regression analysis was applied to assess whether the amount of residual coronal dentin and the type of endocanalar retention had a significant influence on failure risk of the restored teeth.

ELIGIBILITY:
Inclusion Criteria:

* endodontically treated premolars with symptom-free root canal filling and a minimum apical seal of 4 mm, in occlusal function with a natural tooth and in interproximal contact with two adjacent natural teeth.

Exclusion Criteria:

* periapical lesion on the X-ray.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2003-01; Primary Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
survival | 2 years

REFERENCES:
- [Derived] Ferrari M, Sorrentino R, Juloski J, Grandini S, Carrabba M, Discepoli N, Ferrari Cagidiaco E. Post-Retained Single Crowns versus Fixed Dental Prostheses: A 7-Year Prospective Clinical Study. J Dent Res. 2017 Dec;96(13):1490-1497. doi: 10.1177/0022034517724146. Epub 2017 Aug 3. PMID 28771388
- [Derived] Juloski J, Fadda GM, Monticelli F, Fajo-Pascual M, Goracci C, Ferrari M. Four-year Survival of Endodontically Treated Premolars Restored with Fiber Posts. J Dent Res. 2014 Jul;93(7 Suppl):52S-58S. doi: 10.1177/0022034514527970. Epub 2014 Mar 19. PMID 24646637
- [Derived] Ferrari M, Vichi A, Fadda GM, Cagidiaco MC, Tay FR, Breschi L, Polimeni A, Goracci C. A randomized controlled trial of endodontically treated and restored premolars. J Dent Res. 2012 Jul;91(7 Suppl):72S-78S. doi: 10.1177/0022034512447949. PMID 22699672